CLINICAL TRIAL: NCT05530616
Title: Impact of Ultrasound Fetal Weight Estimation on Obstetrical Management and Maternal and Neonatal Outcomes
Acronym: EPF
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8581
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Fetal Weight
Keywords: Fetal Weight; Ultrasound Fetal Weight; Obstetrical Management; Maternal Outcomes; Neonatal Outcomes
MeSH Terms: conditions — Fetal Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators wish to study the obstetrical data of pregnant women who had an ultrasound estimation of fetal weight and who delivered at the University Hospital of Strasbourg over the last 20 years. These retrospectively collected data are a valuable source of scientific information since they are "real life data", currently of growing interest in the scientific community, and have a large volume and quality due to the number of years included and the variety of information collected in the computerized media records.

From this study, the investigators hope not only to better understand the consequences of ultrasound screening for fetal growth, but also to improve its accuracy and to develop useful models in obstetrical decision making in order to decrease maternal and neonatal morbidity.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years of age).
* Female and with a single pregnancy
* Subject having had an ultrasound follow-up at HUS between 01/01/2000 and 31/12/2021
* Subject who gave birth at HUS between 01/01/2000 and 12/31/2021
* Subject who does not object to the reuse of her data for scientific research purposes

Exclusion Criteria:

* Subject who has expressed opposition to the reuse of their data for scientific research purposes
* Multiple pregnancies
* Delivery before 24 weeks of amenorrhea
* Diagnosis of a malformative fetal pathology
* Diagnosis of fetal death in utero

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Major Female (≥18 years of age) with a single pregnancy having had an ultrasound follow-up at HUS between 01/01/2000 and 31/12/2021
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Retrospective study of maternal and neonatal clinical and ultrasound data for the development of an algorithm model useful in obstetrical decision making in order to decrease maternal and neonatal morbidity. | Files analysed retrospectively from January 01, 2000 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - CHU de Strasbourg - France, Strasbourg, France